CLINICAL TRIAL: NCT00929084
Title: Survivor Stories: Impact on Cancer Patients' Quality of Life and Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Donna Jeffe, Professor of Medicine, Director, Health Behavior, Communication and Outreach Core, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 000799
Record Dates: First submitted 2009-06-24; First posted 2009-06-26 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Race Disparities; Breast Cancer; Quality of Life; Treatment Adherence
MeSH Terms: conditions — Breast Neoplasms; Treatment Adherence and Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Survivor Stories Arm (Other): Women in the Survivor Stories intervention arm will be given the Survivor Stories Tablet to take home for two weeks at three different time points over a two year period.
  Interventions: Other: The Survivor Stories Tablet
- Control Arm (Other): Women in the Control Arm will receive standard care.
  Interventions: Other: The Survivor Stories Tablet

INTERVENTIONS:
Other: The Survivor Stories Tablet — The Survivor Stories Tablet is a tablet computer where participants can browse an archive of 1-3 minute videotaped survivor stories told by African American Breast Cancer Survivors. Stories contain five main topics: coping, relationships, experiences with the health care system, follow-up care, and quality of life (QOL) living with breast cancer.

SUMMARY:
The purpose of this study is to evaluate in a randomized controlled trail, an innovative cancer communication strategy to help African American breast cancer patients cope with a variety of challenges during and after treatment and to better adhere to recommended treatment guidelines and follow-up care.

DETAILED DESCRIPTION:
Disparities in incidence and mortality between African Americans and Caucasians for a number of cancers have been well documented. This study builds on previous work in St. Louis to overcome barriers to access to breast screening, identifying and addressing factors associated with access to care once diagnosed, and factors contributing to delay in diagnosis and completion of therapy. African American breast cancer patients randomly assigned to the intervention arm of the trial will have access to the Survivor Stories Tablet, a tablet computer, on which they will browse an archive of 1-3 minute videotaped survivor stories about five topics: coping, relationships, experiences with the health care system, follow-up care, and quality of life (QOL) living with breast cancer. Patients will have the tablet for two weeks after enrollment in the study, and again at 6 and 12 months. Patients in the control arm will receive usual care.

ELIGIBILITY:
Inclusion Criteria:

* African American women
* First primary ductal carcinoma in situ (DCIS) or stages I, II, or III invasive breast cancer.

Exclusion Criteria:

* Prior DCIS or breast cancer diagnosis
* Stage IV or metastatic breast cancer
* Planned to receive a double mastectomy
* non-English speaking,
* Having known psychiatric or neurologic disorders
* Being cognitively impaired according to weighted error scores on the Orientation-Memory-Concentration Test
* Being unwilling or unable to give consent

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2009-11; Primary Completion 2015-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Determine to what extent African American breast cancer survivor stories affect various aspects of QOL, including depressed mood and concern about recurrence, among African American breast cancer patients following primary treatment. | Outcome measures are assessed at five time points: baseline, one month following primary treatment surgery, 6 months, one year, and two years post surgery.

SECONDARY OUTCOMES:
Determine whether and to what extent African American breast cancer survivor stories affect African American breast cancer patients' adherence to recommended surveillance mammography and prescribed hormone therapy | Outcome measures are assessed at five time points: baseline, one month following primary treatment surgery, 6 months, one year, and two years post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Donna B Jeffe, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Thompson T, Perez M, Kreuter M, Margenthaler J, Colditz G, Jeffe DB. Perceived social support in African American breast cancer patients: Predictors and effects. Soc Sci Med. 2017 Nov;192:134-142. doi: 10.1016/j.socscimed.2017.09.035. Epub 2017 Sep 22. PMID 28965004
- [Result] Thompson T, Perez M, Yan Y, Kreuter MW, Margenthaler JA, Colditz GA, Jeffe DB. Randomized controlled trial of a breast cancer Survivor Stories intervention for African American women. Soc Sci Med. 2021 Feb;270:113663. doi: 10.1016/j.socscimed.2020.113663. Epub 2020 Dec 29. PMID 33454539
- [Result] Perez M, Kreuter MW, Yan Y, Thompson T, Sefko J, Golla B, Margenthaler JA, Colditz G, Jeffe DB. Feasibility and Acceptability of an Interactive Cancer-Communication Video Program Using African American Breast Cancer Survivor Stories. J Health Commun. 2020 Jul 2;25(7):566-575. doi: 10.1080/10810730.2020.1821132. Epub 2020 Oct 13. PMID 33048635
- [Result] Jarvandi S, Perez M, Margenthaler J, Colditz GA, Kreuter MW, Jeffe DB. Improving Lifestyle Behaviors After Breast Cancer Treatment Among African American Women With and Without Diabetes: Role of Health Care Professionals. Ann Behav Med. 2021 Feb 12;55(1):1-13. doi: 10.1093/abm/kaaa020. PMID 32298407
- [Result] Schootman M, Perez M, Schootman JC, Fu Q, McVay A, Margenthaler J, Colditz GA, Kreuter MW, Jeffe DB. Influence of built environment on quality of life changes in African-American patients with non-metastatic breast cancer. Health Place. 2020 May;63:102333. doi: 10.1016/j.healthplace.2020.102333. Epub 2020 May 11. PMID 32543424
- [Derived] Cho B, Perez M, Jeffe DB, Kreuter MW, Margenthaler JA, Colditz GA, Liu Y. Factors associated with initiation and continuation of endocrine therapy in women with hormone receptor-positive breast cancer. BMC Cancer. 2022 Aug 1;22(1):837. doi: 10.1186/s12885-022-09946-x. PMID 35915419